CLINICAL TRIAL: NCT05227261
Title: Assessment of a Novel Blood Test in Early Detection of the Five Common Cancers Based on the Investigation of the Circulating Tumour DNA
Brief Title: Early Detection of Five Common Cancers Using the ctDNA Analysing Test
Acronym: K-DETEK
Status: Completed | Type: Observational
Sponsor: Gene Solutions (Industry)
Collaborators: Medical University of Ho Chi Minh City (Unknown); Hanoi Medical University (Other); Hanoi Oncology Hospital (Unknown); Hue Central Hospital (Other); Da Nang Oncology Hospital (Unknown); Thong Nhat Dong Nai General Hospital (Unknown); Dong Nai General Hospital (Unknown); Van Hanh General Hospital (Other); Can Tho Oncology Hospital (Unknown); Medic Medical Center (Unknown); Le Van Thinh Hospital (Other Government); People's Hospital 115 (Unknown); Xuyen A Hospital (Unknown); Medical Genetics Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: 02GS
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Cancer, Lung; Cancer, Breast; Cancer Liver; Cancer, Colorectal; Liquid Biopsy; Circulating Tumour DNA; Cancer, Gastric
Keywords: Early cancer detection; Circulating Tumour DNA; Liquid biopsy; Vietnam
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Carcinoma, Hepatocellular; Colorectal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples collected from the participants will be processed and analysed the ctDNA to detect cancer in the early stages and to predict the origin of the tumor. The residual blood of this test will be stored in -80 degree of Celcius for further testing to:- (i) screen or diagnose cancers; (ii) determine the hosts' genetic factors associated with the risks of cancers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-centre, prospective cohort study, aiming to evaluate a blood test in early detection of the four common cancers, based on the investigation of the circulating tumour DNA (ctDNA).

Primary objective: To evaluate the performance characteristics of the blood ctDNA test in early detecting cancers.

Secondary objectives:

* To evaluate the performance characteristics of the test in determining the origin of tumour, as compared to the findings of the imaging diagnostic tests.
* To determine the risk of cancers development in the high-risk population, as compared to that in the moderate-risk group.

DETAILED DESCRIPTION:
This is a multi-centre, prospective cohort study recruiting participants aged 40 or above, who present at the Outpatient Clinic of the study hospitals either for periodically follow-up visits for their chronic conditions, or for annually health check-up. The study will be conducted at the Medical Genetic Institute, in collaboration with the University of Medicine and Pharmacy at Ho Chi Minh City, Vietnam and other collaborating hospitals.

The potential participants, who satisfy all inclusion/exclusion criteria will be recruited into this study. These potential participants should not have history of cancer before being enrolled in the study.

At enrolment, each participant will answer to a pre-designed questionnaire to provide demographic information, past major medical history and clinical warning signs of cancers, and then provide 10mL of blood for analysing the circulating tumour DNA (ctDNA).

Each participant will get either ctDNA detected or ctDNA not detected.

For those having ctDNA detected in their blood, they will then undergo the screening and diagnostic tests for cancers based on the prediction of tumour origin provided in the test findings report. If the cancers lab-confirmed, patients will then be followed up and managed for their disease according to the guidelines of the Vietnam Ministry of Health and/or the international guidelines on cancers. At 12 months (+/- 1 week) following the enrolment, these patients will be contacted to collect information about their health, in general and their cancer status, in particular.

For those having ctDNA detected in their blood but the present of a mass inside participants' body could not be detected using the imaging diagnostic tests; and for those, who don't have ctDNA presenting in blood, phone calls will be made at 6 months (+/- 1 week) and 12 months (+/- 1 week) following the enrolment to collect information related to participants' health status as well as cancer progress (if possible).

The enrolment is anticipated to last for approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 or above at enrolment
* Neither clinical suspicion of cancer nor history of confirmed cancer has been reported
* Agree to be contacted at 6 months and 12 months following enrolment to collect information about general health status and progress of cancer (if possible)
* Provide written informed consent

Exclusion Criteria: If a potential participant has any one of the following criteria, he/she will not be able to be enrolled in the study:

* History of cancer (cancer has either been confirmed or been treated within the past 3 years)
* History of blood transfusion or bone marrow transplantation within the past 3 years
* Does not agree to participate in study
* The subject has clinical manifestations of pregnant.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include both males and females, aged 40 or above, who have no history of cancer. These people present at the Outpatient Clinic of the study hospitals either for periodically follow-up visits for their chronic conditions or for health check-up.The eligible participants will have to satisfy all of the inclusion and exclusion criteria to be recruited into this study.
Sampling Method: Non-Probability Sample
Enrollment: 9057 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Positive predictive value, Negative predictive value of the blood ctDNA test in early detecting cancers | 12 months following enrolment
Sensitivity and specificity of the test in early detecting cancers | 12 months following enrolment

SECONDARY OUTCOMES:
Positive predictive value of the test in determining the origin of tumour, as compared to the findings of the imaging diagnostic tests | 12 months following enrolment
Rate of cancer development in the high-risk group as compared to the moderate-risk population | 12 months following enrolment

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi medical university, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data of this study may be requested for publication by journals. Sharing anonymised data with future similar/suitable studies will be decided by the sponsor, PIs and the authority agency where the data was collected. No identifiable information will be shared with any other person/organisation than authorized in the study.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Pham T, Bui L, Kim G, Hoang D, Tran T, Hoang M. Cancers in Vietnam-Burden and Control Efforts: A Narrative Scoping Review. Cancer Control. 2019 Jan-Dec;26(1):1073274819863802. doi: 10.1177/1073274819863802. PMID 31319695
- [Background] Ahlquist DA. Universal cancer screening: revolutionary, rational, and realizable. NPJ Precis Oncol. 2018 Oct 29;2:23. doi: 10.1038/s41698-018-0066-x. eCollection 2018. PMID 30393772
- [Background] Brenner H, Jansen L, Ulrich A, Chang-Claude J, Hoffmeister M. Survival of patients with symptom- and screening-detected colorectal cancer. Oncotarget. 2016 Jul 12;7(28):44695-44704. doi: 10.18632/oncotarget.9412. PMID 27213584
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Tabar L, Fagerberg G, Chen HH, Duffy SW, Smart CR, Gad A, Smith RA. Efficacy of breast cancer screening by age. New results from the Swedish Two-County Trial. Cancer. 1995 May 15;75(10):2507-17. doi: 10.1002/1097-0142(19950515)75:103.0.co;2-h. PMID 7736395
- [Background] Cappell MS. The pathophysiology, clinical presentation, and diagnosis of colon cancer and adenomatous polyps. Med Clin North Am. 2005 Jan;89(1):1-42, vii. doi: 10.1016/j.mcna.2004.08.011. PMID 15527807
- [Background] Vahabi M. Breast cancer screening methods: a review of the evidence. Health Care Women Int. 2003 Nov;24(9):773-93. doi: 10.1080/07399330390229957. PMID 14742116
- [Background] Chen X, Gole J, Gore A, He Q, Lu M, Min J, Yuan Z, Yang X, Jiang Y, Zhang T, Suo C, Li X, Cheng L, Zhang Z, Niu H, Li Z, Xie Z, Shi H, Zhang X, Fan M, Wang X, Yang Y, Dang J, McConnell C, Zhang J, Wang J, Yu S, Ye W, Gao Y, Zhang K, Liu R, Jin L. Non-invasive early detection of cancer four years before conventional diagnosis using a blood test. Nat Commun. 2020 Jul 21;11(1):3475. doi: 10.1038/s41467-020-17316-z. PMID 32694610
- [Background] Bradley SH, Kennedy MPT, Neal RD. Recognising Lung Cancer in Primary Care. Adv Ther. 2019 Jan;36(1):19-30. doi: 10.1007/s12325-018-0843-5. Epub 2018 Nov 29. PMID 30499068
- [Background] Hubbell E, Clarke CA, Aravanis AM, Berg CD. Modeled Reductions in Late-stage Cancer with a Multi-Cancer Early Detection Test. Cancer Epidemiol Biomarkers Prev. 2021 Mar;30(3):460-468. doi: 10.1158/1055-9965.EPI-20-1134. Epub 2020 Dec 16. PMID 33328254
- [Background] Simmons C, Milburn J. Impact of Low-Dose Computed Tomography on Computed Tomography Orders and Scan Length. Ochsner J. 2019 Winter;19(4):303-308. doi: 10.31486/toj.19.0008. PMID 31903052
- [Background] Newton KF, Newman W, Hill J. Review of biomarkers in colorectal cancer. Colorectal Dis. 2012 Jan;14(1):3-17. doi: 10.1111/j.1463-1318.2010.02439.x. PMID 21040359
- [Background] Locker GY, Hamilton S, Harris J, Jessup JM, Kemeny N, Macdonald JS, Somerfield MR, Hayes DF, Bast RC Jr; ASCO. ASCO 2006 update of recommendations for the use of tumor markers in gastrointestinal cancer. J Clin Oncol. 2006 Nov 20;24(33):5313-27. doi: 10.1200/JCO.2006.08.2644. Epub 2006 Oct 23. PMID 17060676
- [Background] Hundt S, Haug U, Brenner H. Blood markers for early detection of colorectal cancer: a systematic review. Cancer Epidemiol Biomarkers Prev. 2007 Oct;16(10):1935-53. doi: 10.1158/1055-9965.EPI-06-0994. PMID 17932341
- [Background] Hauptman N, Glavac D. Colorectal Cancer Blood-Based Biomarkers. Gastroenterol Res Pract. 2017;2017:2195361. doi: 10.1155/2017/2195361. Epub 2017 Sep 25. PMID 29147109
- [Background] Church TR, Wandell M, Lofton-Day C, Mongin SJ, Burger M, Payne SR, Castanos-Velez E, Blumenstein BA, Rosch T, Osborn N, Snover D, Day RW, Ransohoff DF; PRESEPT Clinical Study Steering Committee, Investigators and Study Team. Prospective evaluation of methylated SEPT9 in plasma for detection of asymptomatic colorectal cancer. Gut. 2014 Feb;63(2):317-25. doi: 10.1136/gutjnl-2012-304149. Epub 2013 Feb 13. PMID 23408352
- [Background] Clarke CA, Hubbell E, Ofman JJ. Multi-cancer early detection: A new paradigm for reducing cancer-specific and all-cause mortality. Cancer Cell. 2021 Apr 12;39(4):447-448. doi: 10.1016/j.ccell.2021.02.004. Epub 2021 Feb 18. No abstract available. PMID 33606995
- [Background] Cristiano S, Leal A, Phallen J, Fiksel J, Adleff V, Bruhm DC, Jensen SO, Medina JE, Hruban C, White JR, Palsgrove DN, Niknafs N, Anagnostou V, Forde P, Naidoo J, Marrone K, Brahmer J, Woodward BD, Husain H, van Rooijen KL, Orntoft MW, Madsen AH, van de Velde CJH, Verheij M, Cats A, Punt CJA, Vink GR, van Grieken NCT, Koopman M, Fijneman RJA, Johansen JS, Nielsen HJ, Meijer GA, Andersen CL, Scharpf RB, Velculescu VE. Genome-wide cell-free DNA fragmentation in patients with cancer. Nature. 2019 Jun;570(7761):385-389. doi: 10.1038/s41586-019-1272-6. Epub 2019 May 29. PMID 31142840
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] Diehl F, Li M, Dressman D, He Y, Shen D, Szabo S, Diaz LA Jr, Goodman SN, David KA, Juhl H, Kinzler KW, Vogelstein B. Detection and quantification of mutations in the plasma of patients with colorectal tumors. Proc Natl Acad Sci U S A. 2005 Nov 8;102(45):16368-73. doi: 10.1073/pnas.0507904102. Epub 2005 Oct 28. PMID 16258065
- [Background] Diehl F, Schmidt K, Choti MA, Romans K, Goodman S, Li M, Thornton K, Agrawal N, Sokoll L, Szabo SA, Kinzler KW, Vogelstein B, Diaz LA Jr. Circulating mutant DNA to assess tumor dynamics. Nat Med. 2008 Sep;14(9):985-90. doi: 10.1038/nm.1789. Epub 2007 Jul 31. PMID 18670422
- [Background] Durham AL, Adcock IM. The relationship between COPD and lung cancer. Lung Cancer. 2015 Nov;90(2):121-7. doi: 10.1016/j.lungcan.2015.08.017. Epub 2015 Aug 29. PMID 26363803
- [Background] Ferlay J, Colombet M, Soerjomataram I, Parkin DM, Pineros M, Znaor A, Bray F. Cancer statistics for the year 2020: An overview. Int J Cancer. 2021 Apr 5. doi: 10.1002/ijc.33588. Online ahead of print. PMID 33818764
- [Background] Garcia-Murillas I, Schiavon G, Weigelt B, Ng C, Hrebien S, Cutts RJ, Cheang M, Osin P, Nerurkar A, Kozarewa I, Garrido JA, Dowsett M, Reis-Filho JS, Smith IE, Turner NC. Mutation tracking in circulating tumor DNA predicts relapse in early breast cancer. Sci Transl Med. 2015 Aug 26;7(302):302ra133. doi: 10.1126/scitranslmed.aab0021. PMID 26311728
- [Background] Gerlinger M, Rowan AJ, Horswell S, Math M, Larkin J, Endesfelder D, Gronroos E, Martinez P, Matthews N, Stewart A, Tarpey P, Varela I, Phillimore B, Begum S, McDonald NQ, Butler A, Jones D, Raine K, Latimer C, Santos CR, Nohadani M, Eklund AC, Spencer-Dene B, Clark G, Pickering L, Stamp G, Gore M, Szallasi Z, Downward J, Futreal PA, Swanton C. Intratumor heterogeneity and branched evolution revealed by multiregion sequencing. N Engl J Med. 2012 Mar 8;366(10):883-892. doi: 10.1056/NEJMoa1113205. PMID 22397650
- [Background] Colomer R, Ruibal A, Genolla J, Salvador L. Circulating CA 15-3 antigen levels in non-mammary malignancies. Br J Cancer. 1989 Feb;59(2):283-6. doi: 10.1038/bjc.1989.58. PMID 2930693
- [Background] Duffy MJ. Serum tumor markers in breast cancer: are they of clinical value? Clin Chem. 2006 Mar;52(3):345-51. doi: 10.1373/clinchem.2005.059832. Epub 2006 Jan 12. PMID 16410341
- [Background] Park BW, Oh JW, Kim JH, Park SH, Kim KS, Kim JH, Lee KS. Preoperative CA 15-3 and CEA serum levels as predictor for breast cancer outcomes. Ann Oncol. 2008 Apr;19(4):675-81. doi: 10.1093/annonc/mdm538. Epub 2007 Nov 23. PMID 18037623
- [Background] Bray C, Bell LN, Liang H, Collins D, Yale SH. Colorectal Cancer Screening. WMJ. 2017 Feb;116(1):27-33. PMID 29099566
- [Background] Jahr S, Hentze H, Englisch S, Hardt D, Fackelmayer FO, Hesch RD, Knippers R. DNA fragments in the blood plasma of cancer patients: quantitations and evidence for their origin from apoptotic and necrotic cells. Cancer Res. 2001 Feb 15;61(4):1659-65. PMID 11245480
- [Background] Schwarzenbach H, Hoon DS, Pantel K. Cell-free nucleic acids as biomarkers in cancer patients. Nat Rev Cancer. 2011 Jun;11(6):426-37. doi: 10.1038/nrc3066. Epub 2011 May 12. PMID 21562580
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Jiang P, Chan CW, Chan KC, Cheng SH, Wong J, Wong VW, Wong GL, Chan SL, Mok TS, Chan HL, Lai PB, Chiu RW, Lo YM. Lengthening and shortening of plasma DNA in hepatocellular carcinoma patients. Proc Natl Acad Sci U S A. 2015 Mar 17;112(11):E1317-25. doi: 10.1073/pnas.1500076112. Epub 2015 Feb 2. PMID 25646427
- [Background] Underhill HR, Kitzman JO, Hellwig S, Welker NC, Daza R, Baker DN, Gligorich KM, Rostomily RC, Bronner MP, Shendure J. Fragment Length of Circulating Tumor DNA. PLoS Genet. 2016 Jul 18;12(7):e1006162. doi: 10.1371/journal.pgen.1006162. eCollection 2016 Jul. PMID 27428049
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Johnson DA, Barclay RL, Mergener K, Weiss G, Konig T, Beck J, Potter NT. Plasma Septin9 versus fecal immunochemical testing for colorectal cancer screening: a prospective multicenter study. PLoS One. 2014 Jun 5;9(6):e98238. doi: 10.1371/journal.pone.0098238. eCollection 2014. PMID 24901436
- [Background] Xu X, Hou Y, Yin X, Bao L, Tang A, Song L, Li F, Tsang S, Wu K, Wu H, He W, Zeng L, Xing M, Wu R, Jiang H, Liu X, Cao D, Guo G, Hu X, Gui Y, Li Z, Xie W, Sun X, Shi M, Cai Z, Wang B, Zhong M, Li J, Lu Z, Gu N, Zhang X, Goodman L, Bolund L, Wang J, Yang H, Kristiansen K, Dean M, Li Y, Wang J. Single-cell exome sequencing reveals single-nucleotide mutation characteristics of a kidney tumor. Cell. 2012 Mar 2;148(5):886-95. doi: 10.1016/j.cell.2012.02.025. PMID 22385958
- [Background] Lipson EJ, Velculescu VE, Pritchard TS, Sausen M, Pardoll DM, Topalian SL, Diaz LA Jr. Circulating tumor DNA analysis as a real-time method for monitoring tumor burden in melanoma patients undergoing treatment with immune checkpoint blockade. J Immunother Cancer. 2014 Dec 16;2(1):42. doi: 10.1186/s40425-014-0042-0. eCollection 2014. PMID 25516806
- [Background] Tie J, Kinde I, Wang Y, Wong HL, Roebert J, Christie M, Tacey M, Wong R, Singh M, Karapetis CS, Desai J, Tran B, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA as an early marker of therapeutic response in patients with metastatic colorectal cancer. Ann Oncol. 2015 Aug;26(8):1715-22. doi: 10.1093/annonc/mdv177. Epub 2015 Apr 7. PMID 25851626
- [Background] Olsson E, Winter C, George A, Chen Y, Howlin J, Tang MH, Dahlgren M, Schulz R, Grabau D, van Westen D, Ferno M, Ingvar C, Rose C, Bendahl PO, Ryden L, Borg A, Gruvberger-Saal SK, Jernstrom H, Saal LH. Serial monitoring of circulating tumor DNA in patients with primary breast cancer for detection of occult metastatic disease. EMBO Mol Med. 2015 Aug;7(8):1034-47. doi: 10.15252/emmm.201404913. PMID 25987569
- [Background] Newman AM, Bratman SV, To J, Wynne JF, Eclov NC, Modlin LA, Liu CL, Neal JW, Wakelee HA, Merritt RE, Shrager JB, Loo BW Jr, Alizadeh AA, Diehn M. An ultrasensitive method for quantitating circulating tumor DNA with broad patient coverage. Nat Med. 2014 May;20(5):548-54. doi: 10.1038/nm.3519. Epub 2014 Apr 6. PMID 24705333
- [Background] Newman AM, Lovejoy AF, Klass DM, Kurtz DM, Chabon JJ, Scherer F, Stehr H, Liu CL, Bratman SV, Say C, Zhou L, Carter JN, West RB, Sledge GW, Shrager JB, Loo BW Jr, Neal JW, Wakelee HA, Diehn M, Alizadeh AA. Integrated digital error suppression for improved detection of circulating tumor DNA. Nat Biotechnol. 2016 May;34(5):547-555. doi: 10.1038/nbt.3520. Epub 2016 Mar 28. PMID 27018799
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Torre LA, Siegel RL, Jemal A. Lung Cancer Statistics. Adv Exp Med Biol. 2016;893:1-19. doi: 10.1007/978-3-319-24223-1_1. PMID 26667336
- [Background] Zahnd WE, Eberth JM. Lung Cancer Screening Utilization: A Behavioral Risk Factor Surveillance System Analysis. Am J Prev Med. 2019 Aug;57(2):250-255. doi: 10.1016/j.amepre.2019.03.015. Epub 2019 Jun 24. PMID 31248742
- [Background] Kim JJ, Burger EA, Regan C, Sy S. Screening for Cervical Cancer in Primary Care: A Decision Analysis for the US Preventive Services Task Force. JAMA. 2018 Aug 21;320(7):706-714. doi: 10.1001/jama.2017.19872. PMID 30140882
- [Background] Lehman CD, Arao RF, Sprague BL, Lee JM, Buist DS, Kerlikowske K, Henderson LM, Onega T, Tosteson AN, Rauscher GH, Miglioretti DL. National Performance Benchmarks for Modern Screening Digital Mammography: Update from the Breast Cancer Surveillance Consortium. Radiology. 2017 Apr;283(1):49-58. doi: 10.1148/radiol.2016161174. Epub 2016 Dec 5. PMID 27918707
- [Background] Pinsky PF, Gierada DS, Black W, Munden R, Nath H, Aberle D, Kazerooni E. Performance of Lung-RADS in the National Lung Screening Trial: a retrospective assessment. Ann Intern Med. 2015 Apr 7;162(7):485-91. doi: 10.7326/M14-2086. PMID 25664444
- [Background] Ofman JJ, Fendrick AM, Raza A. Novel multicancer early detection technology-potential value to employers and the workforce. Am J Manag Care. 2020 Dec;26(10 Spec No.):SP363. doi: 10.37765/ajmc.2020.88567. PMID 33395237
- [Background] Cohen JD, Li L, Wang Y, Thoburn C, Afsari B, Danilova L, Douville C, Javed AA, Wong F, Mattox A, Hruban RH, Wolfgang CL, Goggins MG, Dal Molin M, Wang TL, Roden R, Klein AP, Ptak J, Dobbyn L, Schaefer J, Silliman N, Popoli M, Vogelstein JT, Browne JD, Schoen RE, Brand RE, Tie J, Gibbs P, Wong HL, Mansfield AS, Jen J, Hanash SM, Falconi M, Allen PJ, Zhou S, Bettegowda C, Diaz LA Jr, Tomasetti C, Kinzler KW, Vogelstein B, Lennon AM, Papadopoulos N. Detection and localization of surgically resectable cancers with a multi-analyte blood test. Science. 2018 Feb 23;359(6378):926-930. doi: 10.1126/science.aar3247. Epub 2018 Jan 18. PMID 29348365
- [Background] Liu MC. Transforming the landscape of early cancer detection using blood tests-Commentary on current methodologies and future prospects. Br J Cancer. 2021 Apr;124(9):1475-1477. doi: 10.1038/s41416-020-01223-7. Epub 2021 Feb 9. PMID 33558712
- [Background] Mathios D, Johansen JS, Cristiano S, Medina JE, Phallen J, Larsen KR, Bruhm DC, Niknafs N, Ferreira L, Adleff V, Chiao JY, Leal A, Noe M, White JR, Arun AS, Hruban C, Annapragada AV, Jensen SO, Orntoft MW, Madsen AH, Carvalho B, de Wit M, Carey J, Dracopoli NC, Maddala T, Fang KC, Hartman AR, Forde PM, Anagnostou V, Brahmer JR, Fijneman RJA, Nielsen HJ, Meijer GA, Andersen CL, Mellemgaard A, Bojesen SE, Scharpf RB, Velculescu VE. Detection and characterization of lung cancer using cell-free DNA fragmentomes. Nat Commun. 2021 Aug 20;12(1):5060. doi: 10.1038/s41467-021-24994-w. PMID 34417454
- [Background] Liu L, Toung JM, Jassowicz AF, Vijayaraghavan R, Kang H, Zhang R, Kruglyak KM, Huang HJ, Hinoue T, Shen H, Salathia NS, Hong DS, Naing A, Subbiah V, Piha-Paul SA, Bibikova M, Granger G, Barnes B, Shen R, Gutekunst K, Fu S, Tsimberidou AM, Lu C, Eng C, Moulder SL, Kopetz ES, Amaria RN, Meric-Bernstam F, Laird PW, Fan JB, Janku F. Targeted methylation sequencing of plasma cell-free DNA for cancer detection and classification. Ann Oncol. 2018 Jun 1;29(6):1445-1453. doi: 10.1093/annonc/mdy119. PMID 29635542
- [Background] Liu MC, Oxnard GR, Klein EA, Swanton C, Seiden MV; CCGA Consortium. Sensitive and specific multi-cancer detection and localization using methylation signatures in cell-free DNA. Ann Oncol. 2020 Jun;31(6):745-759. doi: 10.1016/j.annonc.2020.02.011. Epub 2020 Mar 30. PMID 33506766
- [Background] Dang AH, Tran VU, Tran TT, Thi Pham HA, Le DT, Nguyen L, Nguyen NV, Thi Nguyen TH, Nguyen CV, Le HT, Thi Nguyen ML, Le VT, Nguyen PH, Vo BT, Thi Dao HT, Nguyen LT, Van Nguyen TC, Bui QN, Nguyen LH, Nguyen NH, Thi Nguyen QT, Le TX, Do TT, Dinh KT, Do HN, Phan MD, Nguyen HN, Tran LS, Giang H. Actionable Mutation Profiles of Non-Small Cell Lung Cancer patients from Vietnamese population. Sci Rep. 2020 Feb 17;10(1):2707. doi: 10.1038/s41598-020-59744-3. PMID 32066856
- [Background] Nguyen HN, Cao NT, Van Nguyen TC, Le KND, Nguyen DT, Nguyen QT, Nguyen TT, Van Nguyen C, Le HT, Nguyen MT, Nguyen TV, Tran VU, Luong BA, Le LGH, Ho QC, Pham HT, Vo BT, Nguyen LT, Dang AH, Nguyen SD, Do DM, Do TT, Hoang AV, Dinh KT, Phan MD, Giang H, Tran LS. Liquid biopsy uncovers distinct patterns of DNA methylation and copy number changes in NSCLC patients with different EGFR-TKI resistant mutations. Sci Rep. 2021 Aug 12;11(1):16436. doi: 10.1038/s41598-021-95985-6. PMID 34385540
- [Background] Nguyen HT, Tran DH, Ngo QD, Pham HT, Tran TT, Tran VU, Pham TN, Le TK, Le NT, Nguyen NM, Vo BT, Nguyen LT, Nguyen TV, Bui QTN, Nguyen HN, Luong BA, Le LGH, Do DM, Do TT, Hoang AV, Dinh KT, Phan MD, Tran LS, Giang H, Nguyen HN. Evaluation of a Liquid Biopsy Protocol using Ultra-Deep Massive Parallel Sequencing for Detecting and Quantifying Circulation Tumor DNA in Colorectal Cancer Patients. Cancer Invest. 2020 Feb;38(2):85-93. doi: 10.1080/07357907.2020.1713350. Epub 2020 Jan 24. PMID 31939681
- [Background] Tran LS, Nguyen QT, Nguyen CV, Tran VU, Nguyen TT, Le HT, Nguyen MT, Le VT, Pham LS, Vo BT, Dang AH, Nguyen LT, Nguyen TV, Pham HT, Tran TT, Nguyen LH, Nguyen TT, Nguyen KT, Vu YV, Nguyen NH, Bui VQ, Bui HH, Do TT, Lam NV, Truong Dinh K, Phan MD, Nguyen HN, Giang H. Ultra-Deep Massive Parallel Sequencing of Plasma Cell-Free DNA Enables Large-Scale Profiling of Driver Mutations in Vietnamese Patients With Advanced Non-Small Cell Lung Cancer. Front Oncol. 2020 Aug 4;10:1351. doi: 10.3389/fonc.2020.01351. eCollection 2020. PMID 32850431
- [Background] Tran LS, Pham HT, Tran VU, Tran TT, Dang AH, Le DT, Nguyen SL, Nguyen NV, Nguyen TV, Vo BT, Dao HT, Nguyen NH, Tran TH, Nguyen CV, Pham PC, Dang-Mai AT, Dinh-Nguyen TK, Phan VH, Do TT, Truong Dinh K, Do HN, Phan MD, Giang H, Nguyen HN. Ultra-deep massively parallel sequencing with unique molecular identifier tagging achieves comparable performance to droplet digital PCR for detection and quantification of circulating tumor DNA from lung cancer patients. PLoS One. 2019 Dec 16;14(12):e0226193. doi: 10.1371/journal.pone.0226193. eCollection 2019. PMID 31841547
- [Background] Lo YMD, Han DSC, Jiang P, Chiu RWK. Epigenetics, fragmentomics, and topology of cell-free DNA in liquid biopsies. Science. 2021 Apr 9;372(6538):eaaw3616. doi: 10.1126/science.aaw3616. PMID 33833097
- [Background] US Preventive Services Task Force; Krist AH, Davidson KW, Mangione CM, Barry MJ, Cabana M, Caughey AB, Davis EM, Donahue KE, Doubeni CA, Kubik M, Landefeld CS, Li L, Ogedegbe G, Owens DK, Pbert L, Silverstein M, Stevermer J, Tseng CW, Wong JB. Screening for Lung Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2021 Mar 9;325(10):962-970. doi: 10.1001/jama.2021.1117. PMID 33687470
- [Derived] Nguyen LHD, Nguyen THH, Le VH, Bui VQ, Nguyen LH, Pham NH, Phan TH, Nguyen HT, Tran VS, Bui CV, Vo VK, Nguyen PTN, Dang HHP, Pham VD, Cao VT, Phan NM, Tieu BL, Nguyen GTH, Vo DH, Tran TH, Nguyen TD, Nguyen VTC, Nguyen TH, Tran VU, Le MP, Tran TMT, Nguyen Nguyen M, Van TTV, Nguyen AN, Nguyen TT, Doan NNT, Nguyen HT, Doan PL, Huynh LAK, Nguyen TA, Nguyen HTP, Lu YT, Cao CTT, Nguyen VT, Le Quyen Le T, Luong TL, Doan TKP, Dao TT, Phan CD, Nguyen TX, Pham NT, Nguyen BT, Pham TTT, Le HL, Truong CT, Jasmine TX, Le MC, Phan VB, Truong QB, Tran THL, Huynh MT, Tran TQ, Nguyen ST, Tran V, Tran VK, Nguyen Nguyen H, Nguyen DS, Van Phan T, Do TT, Truong DK, Tang HS, Giang H, Nguyen HN, Phan MD, Tran LS. Prospective validation study: a non-invasive circulating tumor DNA-based assay for simultaneous early detection of multiple cancers in asymptomatic adults. BMC Med. 2025 Feb 14;23(1):90. doi: 10.1186/s12916-025-03929-y. PMID 39948555
- See also: World Health Organization. Firm action is needed to eliminate viral hepatitis in Viet Nam. 2017 — https://www.who.int/vietnam/news/detail/28-07-2017-firm-action-is-needed-to-eliminate-viral-hepatitis-in-viet-nam
- See also: World Health Organization. Vietnam: International Agency for Research on Cancer. 2021 — https://gco.iarc.fr/today/data/factsheets/populations/704-viet-nam-fact-sheets.pdf